CLINICAL TRIAL: NCT01992094
Title: A Phase III, Stratified, Randomized, Double-Blind, Multicenter, NonInferiority Study to Evaluate the Safety and Immunogenicity of a Cell-based Quadrivalent Subunit Influenza Virus Vaccine and Cell-based Trivalent Subunit Influenza Virus Vaccines in Adults Ages ≥18 Years of Age
Brief Title: Safety and Immunogenicity of Three Influenza Vaccines Adults Ages 18 and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V130_01
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Influenza
Keywords: Influenza; Influenza vaccine; Novartis; Adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- QIVc (Experimental): Influenza vaccine
  Interventions: Biological: QIVc
- TIV1c (Active Comparator): Influenza vaccine
  Interventions: Biological: TIV1c
- TIV2c (Active Comparator): Influenza vaccine
  Interventions: Biological: TIV2c

INTERVENTIONS:
Biological: QIVc — Novartis Investigational Quadrivalent Vaccine
  Arms: QIVc
Biological: TIV1c — Licensed Influenza Vaccine
  Arms: TIV1c
Biological: TIV2c — Novartis Investigational Vaccine
  Arms: TIV2c

SUMMARY:
Evaluate safety and immunogenicity of three influenza vaccines in adults 18 years of age and above.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 18 years and older.
2. Individuals who give written informed consent, who can comply with study procedures, and who are available for follow-up.

Exclusion Criteria:

1. Individuals recently vaccinated against influenza
2. Subjects with contraindications to receive influenza vaccine
3. Please contact the site for additional eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2680 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (36):
- United States (36):
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Anaheim, California
  - San Diego, California
  - Coral Gables, Florida
  - Hollywood, Florida
  - Melbourne, Florida
  - South Miami, Florida
  - West Palm Beach, Florida
  - Peoria, Illinois
  - Mishawaka, Indiana
  - Council Bluffs, Iowa
  - Newton, Kansas
  - Wichita, Kansas
  - Metairie, Louisiana
  - Rockville, Maryland
  - Edina, Minnesota
  - Bellevue, Nebraska
  - Omaha, Nebraska
  - Endwell, New York
  - Rochester, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Oklahoma City, Oklahoma
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Mt. Pleasant, South Carolina
  - Dakota Dunes, South Dakota
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Salt Lake City, Utah
  - South Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 40 centers in US
Pre-assignment Details: All enrolled subjects were included in the trial
Groups:
- QIVc (≥18 Years): Subjects received one dose of cell derived quadrivalent influenza vaccine (QIVc)
- TIV1c (≥18 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV1c (H1N1,H3N2, B1) recommended for 2013-2014 season
- TIV2c (≥18 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV2c that contains an alternate B strain compared to what is recommended for 2013-2014
Period: Overall Study
Arm/Group | QIVc (≥18 Years) | TIV1c (≥18 Years) | TIV2c (≥18 Years)
Started | 1335 | 676 | 669
Completed | 1285 | 652 | 648
Not Completed | 50 | 24 | 21
Not completed — ADMINISTRATIVE REASON | 6 | 7 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 5 | 5 | 2
Not completed — Lost to Follow-up | 26 | 9 | 13
Not completed — OTHER | 4 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QIVc (≥18 Years) | TIV1c (≥18 Years) | TIV2c (≥18 Years) | Total
Number analyzed (Participants) | 1335 | 676 | 669 | 2680
Age, Continuous [Mean (Standard Deviation); unit: year] | 57.4 (17.8) | 57.2 (18.0) | 57.1 (18.1) | 57.3 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 732 | 392 | 392 | 1516
  Male | 603 | 284 | 277 | 1164

OUTCOME MEASURES:

1. Primary Outcome: 1.Geometric Mean Titres (GMT) in Subjects After Receiving One Dose of Either QIVc, TIV1c or TIV2c
Description: Immunogenicity of QIVc to comparator TIVc (For H1N1, H3N2 and B1 strain, the comparison is between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison is between QIVc and TIV2c) was assessed in terms of GMT in subjects measured by hemagglutination inhibition (HI) assay, three weeks after vaccination with one dose of either QIVc or TIV1c and TIV2c.
  Non-inferiority was established if the upper bound of the two-sided 95% confidence interval (CI) for the ratio of GMTs (GMT TIV1c or TIV2c /GMT QIVc) for HI antibody does not exceed the non-inferiority margin of 1.5.
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on Per Protocol (PP) Population i.e. all subjects in the Full Analysis Set (FAS) efficacy/immunogenicity population correctly receive the vaccine, have no major protocol deviations leading to exclusion as defined prior to unblinding/analysis and are not excluded due to other reasons defined prior to unblinding or analysis
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- TIV1c (≥18 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV1c (H1N1, H3N2, B1) recommended for 2013-2014 season
Arm/Group | QIVc (≥18 Years) | TIV1c (≥18 Years) | TIV2c (≥18 Years)
Number analyzed (Participants) | 1335 | 676 | 669
Titer
  H1N1: Day 1(N=1250,635,NA) | 60.7 [56.0 to 65.9] | 59.6 [53.0 to 67.0] | NA [NA to NA] — antigen not immunized
  H1N1: Day 22(N=1250,635,NA) | 302.8 [281.8 to 325.5] | 298.9 [270.3 to 330.5] | NA [NA to NA] — antigen not immunized
  H3N2: Day 1(N=1250,635,NA) | 122.5 [112.7 to 133.1] | 128.1 [113.6 to 144.6] | NA [NA to NA] — antigen not immunized
  H3N2: Day 22(N=1250,635,NA) | 372.3 [349.2 to 396.9] | 378.4 [345.1 to 414.8] | NA [NA to NA] — antigen not immunized
  B1:Day 1(N=1250,635,NA) | 45.3 [42.6 to 48.1] | 43.8 [40.2 to 47.7] | NA [NA to NA] — antigen not immunized
  B1:Day 22(N=1250,635,NA) | 133.2 [125.3 to 141.7] | 115.6 [106.4 to 125.6] | NA [NA to NA] — antigen not immunized
  B2:Day 1(N=1250,NA,639) | 59.2 [56.0 to 62.7] | NA [NA to NA] — antigen not immunized | 58.0 [53.4 to 63.0]
  B2:Day 22(N=1250,NA,639) | 177.2 [167.6 to 187.5] | NA [NA to NA] — antigen not immunized | 164.0 [151.4 to 177.7]
Statistical Analysis 1: Comparison: QIVc (≥18 Years) vs TIV1c (≥18 Years); Non-inferiority of immune responses of QIVc to TIV1c, assessed in terms of ratios of GMT against influenza strain H1N1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper bound of the two-sided 95% confidence interval (CI) for the ratio of GMTs (GMT TIV1c/GMT QIVc) for HI antibody does not exceed the non-inferiority margin of 1.5; ANCOVA; Ratios of GMT = 1.0, 95% CI 2-sided [0.9 to 1.1]
Statistical Analysis 2: Comparison: QIVc (≥18 Years) vs TIV1c (≥18 Years); Non-inferiority of immune responses of QIVc to TIV1c, assessed in terms of ratios of GMT against influenza strain H3N2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratios of GMT = 1.0, 95% CI 2-sided [0.9 to 1.1]
Statistical Analysis 3: Comparison: QIVc (≥18 Years) vs TIV1c (≥18 Years); Non-inferiority of immune responses of QIVc to TIV1c, assessed in terms of ratios of GMT against influenza strain B1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratios of GMT = 0.9, 95% CI 2-sided [0.8 to 1.0]
Statistical Analysis 4: Comparison: QIVc (≥18 Years) vs TIV2c (≥18 Years); Non-inferiority of immune responses of QIVc to TIV2c, assessed in terms of ratios of GMT against influenza strain B2; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper bound of the two-sided 95% confidence interval (CI) for the ratio of GMTs (GMT TIV2c/GMT QIVc) for HI antibody does not exceed the non-inferiority margin of 1.5; ANCOVA; Ratios of GMT = 0.9, 95% CI 2-sided [0.9 to 1.0]

2. Primary Outcome: 2. Percentages of Subjects Achieving Seroconversion After One Dose of Either QIVc, TIV1c or TIV2c
Description: Immunogenicity of QIVc to comparator TIVc (For H1N1, H3N2 and B1 strain, the comparison is between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison is between QIVc and TIV2c) was assessed in terms of percentages of subjects showing seroconversion or significant increase in HI antibody titers, three weeks (day 22) after vaccination with one dose of either QIVc,TIV1c or TIV2c Seroconversion is defined in subjects seronegative at baseline (i.e., HI titer <1:10 at Day 1) as post-vaccination HI titer ≥1:40, and defined in subjects sero-positive at baseline (i.e., HI titer ≥1:10 at Day 1) as a minimum of a 4-fold increase in post-vaccination HI titer
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on PP population
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | QIVc (≥18 Years) | TIV1c (≥18 Years) | TIV2c (≥18 Years)
Number analyzed (Participants) | 1335 | 676 | 669
percentage of subjects
  H1N1: Day 22(N=1250, 635,NA) | 49.2 [46.4 to 52.0] | 48.7 [44.7 to 52.6] | NA [NA to NA] — antigen not immunized
  H3N2: Day 22(N=1250, 635,NA) | 38.3 [35.6 to 41.1] | 35.6 [31.9 to 39.5] | NA [NA to NA] — antigen not immunized
  B1: Day 22(N=1250, 635,NA) | 36.6 [33.9 to 39.3] | 34.8 [31.1 to 38.7] | NA [NA to NA] — antigen not immunized
  B2: Day 22(N=1250,NA, 639) | 39.8 [37.0 to 42.5] | NA [NA to NA] — antigen not immunized | 35.4 [31.7 to 39.2]
Statistical Analysis 1: Comparison: QIVc (≥18 Years) vs TIV1c (≥18 Years); Non-inferiority of immune responses of QIVc to TIV1c in terms of differences in seroconversion rates against influenza strain H1N1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper bound of the two-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV1c - % seroconversion QIVc) for HI antibody does not exceed the margin of 10%; ANCOVA; Difference between seroconversion rates = -0.5, 95% CI 2-sided [-5.3 to 4.2]
Statistical Analysis 2: Comparison: QIVc (≥18 Years) vs TIV1c (≥18 Years); Non-inferiority of immune responses of QIVc to TIV1c in terms of differences in seroconversion rates against influenza strainH3N2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Difference between seroconversion rates = -2.7, 95% CI 2-sided [-7.2 to 1.9]
Statistical Analysis 3: Comparison: QIVc (≥18 Years) vs TIV1c (≥18 Years); Non-inferiority of immune responses of QIVc to TIV1c in terms of differences in seroconversion rates against influenza strain B1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Difference between seroconversion rates = -1.8, 95% CI 2-sided [-6.2 to 2.8]
Statistical Analysis 4: Comparison: QIVc (≥18 Years) vs TIV2c (≥18 Years); Non-inferiority of immune responses of QIVc to TIV2c in terms of differences in seroconversion rates against influenza strain B2; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper bound of the two-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV2c - % seroconversion QIVc) for HI antibody does not exceed the margin of 10%; ANCOVA; Difference between seroconversion rates = -4.4, 95% CI 2-sided [-8.9 to 0.2]

3. Secondary Outcome: 3. Percentages of Subjects Achieving Seroconversion After One Dose of Either QIVc, TIV1c or TIV2c in 18 to <65 and ≥ 65 Years Age Cohorts
Description: Immunogenicity was assessed in terms of percentages of subjects showing seroconversion or significant increase in HI antibody titers, against each vaccine strains, three weeks (day 22) after vaccination with ether QIVc, TIV1c or TIV2c Seroconversion is defined in subjects seronegative at baseline (i.e., HI titer <1:10 at Day 1) as post-vaccination HI titer ≥1:40, and defined in subjects sero-positive at baseline (i.e., HI titer ≥1:10 at Day 1) as a minimum of a 4-fold increase in post-vaccination HI titer.The CBER criterion for 18 to <65 years age group is that the lower bound of the two-sided 95% CI for the percentage of subjects achieving seroconversion for HI antibody should meet or exceed 40% and that for the ≥ 65 years age group should meet or exceed 30%
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS immunogenicity set i.e. all subjects in the enrolled set who receive the study vaccination and provide immunogenicity data at visit 1 and visit 2
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- QIVc (18 to <65 Years); QIVc (≥ 65 Years): Subjects received one dose of cell derived quadrivalent influenza vaccine (QIVc)
- TIV1c (18 to <65 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV1c (H1N1, H3N2, B1) recommended for 2013- 2014 season
- TIV1c (≥ 65 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV1c (H1N1,H3N2, B1)recommended for 2013-2014 season
- TIV2c (18 to <65 Years); TIV2c (≥ 65 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV2c that contains an alternate B strain compared to what is recommended for 2013-2014
Arm/Group | QIVc (18 to <65 Years) | QIVc (≥ 65 Years) | TIV1c (18 to <65 Years) | TIV1c (≥ 65 Years) | TIV2c (18 to <65 Years) | TIV2c (≥ 65 Years)
Number analyzed (Participants) | 661 | 650 | 328 | 336 | 326 | 332
percentages of subjects
  H1N1: Day 22(N=661, 650, 328, 336,NA,NA) | 63.1 [59.3 to 66.8] | 34.5 [30.8 to 38.3] | 60.4 [54.8 to 65.7] | 36.9 [31.7 to 42.3] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  H3N2: Day 22(N=661, 650, 328, 336,NA,NA) | 49.2 [45.3 to 53.1] | 27.2 [23.8 to 30.8] | 47.3 [41.7 to 52.8] | 24.7 [20.2 to 29.7] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B1: Day 22(N=661, 650, 328, 336,NA,NA) | 52.0 [48.2 to 55.9] | 20.9 [17.9 to 24.3] | 50.3 [44.8 to 55.8] | 19.3 [15.3 to 24.0] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B2: Day 22(N=661, 650,NA,NA, 326, 332) | 52.8 [48.9 to 56.7] | 26.3 [23.0 to 29.9] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized | 50.3 [44.7 to 55.9] | 20.8 [16.5 to 25.6]

4. Secondary Outcome: 4. Percentages of Subjects Achieving HI Titer ≥1:40 After One Dose of Either QIVc, TIV1c or TIV2c in 18 to <65 and ≥ 65 Years Age-cohorts
Description: Immunogenicity was assessed in terms of percentages of subjects showing HI titer ≥1:40, three weeks (day 22) after vaccination with either QIVc, TIV1c or TIV2c The CBER criterion for 18 to <65 years age group is that the lower bound of the two-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥ 1:40 should meet or exceed 70% and that for the ≥ 65 years age group should meet or exceed 60%
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS immunogenicity set.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- TIV1c (18 to <65 Years); TIV1c (≥ 65 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV1c (H1N1,H3N2, B1) recommended for 2013-2014 season
Arm/Group | QIVc (18 to <65 Years) | QIVc (≥ 65 Years) | TIV1c (18 to <65 Years) | TIV1c (≥ 65 Years) | TIV2c (18 to <65 Years) | TIV2c (≥ 65 Years)
Number analyzed (Participants) | 661 | 650 | 328 | 336 | 326 | 332
percentages of subjects
  H1N1: Day 1(N=661, 650, 328, 336,NA,NA) | 63.8 [60.0 to 67.5] | 79.2 [75.9 to 82.3] | 64.6 [59.2 to 69.8] | 76.5 [71.6 to 80.9] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  H1N1: Day 22(N=661, 650, 328, 336,NA,NA) | 98.5 [97.2 to 99.3] | 94.3 [92.2 to 96.0] | 97.0 [94.5 to 98.5] | 96.1 [93.5 to 97.9] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  H3N2: Day 1(N=661, 650, 328, 336,NA,NA) | 78.2 [74.9 to 81.3] | 89.5 [86.9 to 91.8] | 80.5 [75.8 to 84.6] | 88.4 [84.5 to 91.6] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  H3N2: Day 22(N=661, 650, 328, 336,NA,NA) | 98.6 [97.4 to 99.4] | 98.3 [97.0 to 99.2] | 99.1 [97.4 to 99.8] | 98.2 [96.2 to 99.3] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B1: Day 1(N=661, 650, 328, 336,NA,NA) | 64.6 [60.8 to 68.2] | 72.3 [68.7 to 75.7] | 62.8 [57.3 to 68.1] | 67.9 [62.6 to 72.8] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B1: Day 22(N=661, 650, 328, 336,NA,NA) | 95.6 [93.8 to 97.0] | 92.2 [89.8 to 94.1] | 95.7 [92.9 to 97.6] | 87.8 [83.8 to 91.1] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B2: Day 1(N=661, 650,NA,NA, 326, 332) | 74.9 [71.4 to 78.2] | 81.2 [78.0 to 84.2] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized | 73.3 [68.2 to 78.0] | 81.0 [76.4 to 85.1]
  B2: Day 22(N=661, 650,NA,NA, 326, 332) | 99.1 [98.0 to 99.7] | 96.2 [94.4 to 97.5] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized | 98.8 [96.9 to 99.7] | 95.2 [92.3 to 97.2]

5. Secondary Outcome: 5.Geometric Mean Ratios (GMR) in Subjects After One Dose of Either QIVc, TIV1c or TIV2c in 18 to ≤60 Years and ≥ 61 Years Age Cohorts
Description: Immunogenicity was measured as the geometric mean ratio (GMR). The ratio of post-vaccination to pre-vaccination HI GMTs, three weeks (day 22) after vaccination with either QIVc, TIV1c or TIV2c Committee for Medicinal Products for Human Use (CHMP) criterion for 18 to ≤60 years age group is >2.5 and that for ≥ 61 years age group is >2.0
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS immunogenicity set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- QIVc (18 to ≤60 Years); QIVc (≥ 61 Years): Subjects received one dose of cell derived quadrivalent influenza vaccine (QIVc)
- TIV1c (18 to ≤60 Years); TIV1c (≥ 61 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV1c (H1N1,H3N2, B1) recommended for 2013- 2014 season
- TIV2c (18 to ≤60 Years); TIV2c (≥ 61 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV2c that contains an alternate B strain compared to what is recommended for 2013-2014
Arm/Group | QIVc (18 to ≤60 Years) | QIVc (≥ 61 Years) | TIV1c (18 to ≤60 Years) | TIV1c (≥ 61 Years) | TIV2c (18 to ≤60 Years) | TIV2c (≥ 61 Years)
Number analyzed (Participants) | 606 | 705 | 306 | 358 | 297 | 361
Ratio
  A/H1N1(Day 22/Day1)(N=606,705,306,358,NA,NA) | 9.2 [8.0 to 10.6] | 3.0 [2.7 to 3.2] | 9.1 [7.5 to 11.1] | 3.0 [2.7 to 3.4] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  A/H3N2 (Day 22/Day1)(N=606,705,306,358,NA,NA) | 4.2 [3.8 to 4.7] | 2.3 [2.1 to 2.5] | 4.2 [3.6 to 4.9] | 2.2 [2.0 to 2.5] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B1 (Day 22/Day1)(N=606,705,306,358,NA,NA) | 4.5 [4.0 to 5.0] | 2.1 [1.9 to 2.2] | 4.1 [3.5 to 4.8] | 1.8 [1.7 to 2.0] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B2 (Day 22/Day1)(N=606,705,NA,NA,297,361) | 4.3 [3.9 to 4.8] | 2.2 [2.0 to 2.3] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized | 4.1 [3.5 to 4.7] | 2.1 [1.9 to 2.3]

6. Secondary Outcome: 6. Percentages of Subjects Achieving Seroconversion After One Dose of Either QIVc, TIV1c or TIV2c in 18 to ≤60 Years and ≥ 61 Years Age Cohorts
Description: Immunogenicity was assessed in terms of percentages of subjects showing seroconversion or significant increase in HI antibody titers, three weeks (day 22) after vaccination with either QIVc, TIV1c or TIV2c Seroconversion is defined in subjects seronegative at baseline (i.e., HI titer <1:10 at Day 1) as post-vaccination HI titer ≥1:40, and defined in subjects sero-positive at baseline (i.e., HI titer ≥1:10 at Day 1) as a minimum of a 4-fold increase in post-vaccination HI titer The CHMP criterion for 18 to ≤60 years age group is that the percentage of subjects achieving seroconversion or significant increase in HI titer is >40% and that for ≥ 61 years age group is >30%
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS immunogenicity set.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (18 to ≤60 Years) | QIVc (≥ 61 Years) | TIV1c (18 to ≤60 Years) | TIV1c (≥ 61 Years) | TIV2c (18 to ≤60 Years) | TIV2c (≥ 61 Years)
Number analyzed (Participants) | 606 | 705 | 306 | 358 | 297 | 361
percentages of subjects
  H1N1: Day 22(N=606,705,306,358,NA,NA) | 63.5 [59.6 to 67.4] | 36.3 [32.8 to 40.4] | 62.1 [56.4 to 67.6] | 36.9 [31.9 to 42.1] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  H3N2: Day 22(N=606,705,306,358,NA,NA) | 49.8 [45.8 to 53.9] | 28.4 [25.1 to 31.9] | 48.7 [43.0 to 54.4] | 24.9 [20.5 to 29.7] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B1: Day 22(N=606,705,306,358,NA,NA) | 53.3 [49.2 to 57.3] | 22.3 [19.2 to 25.5] | 52.3 [46.5 to 58.0] | 19.6 [15.6 to 24.0] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B2: Day 22(N=606,705,NA,NA,297,361) | 53.8 [49.7 to 57.8] | 27.5 [24.3 to 31.0] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized | 51.2 [45.3 to 57.0] | 22.4 [18.2 to 27.1]

7. Secondary Outcome: 7. Percentages of Subjects Achieving HI Titer ≥1:40 After One Dose of Either QIVc, TIV1c or TIV2c in 18 to ≤60 Years and ≥ 61 Years Age Cohorts
Description: Immunogenicity was assessed in terms of percentages of subjects showing HI titer ≥1:40, three weeks (day 22) after vaccination with either QIVc, TIV1c and TIV2c The CHMP criterion for 18 to ≤60 years age group is that the percentage of subjects achieving an HI titer ≥1:40 is >70% and that for ≥ 61 years age group is >60%
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS immunogenicity set.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (18 to ≤60 Years) | QIVc (≥ 61 Years) | TIV1c (18 to ≤60 Years) | TIV1c (≥ 61 Years) | TIV2c (18 to ≤60 Years) | TIV2c (≥ 61 Years)
Number analyzed (Participants) | 606 | 705 | 306 | 358 | 297 | 361
percentages of subjects
  H1N1: Day 1(N=606,705,306,358,NA,NA) | 64.4 [60.4 to 68.2] | 77.6 [74.3 to 80.6] | 65.0 [59.4 to 70.4] | 75.4 [70.6 to 79.8] | NA [NA to NA] — antigen not immunized | NA [0 to 0] — antigen not immunized
  H1N1: Day 22(N=606,705,306,358,NA,NA) | 98.3 [97.0 to 99.2] | 94.8 [92.8 to 96.3] | 97.4 [94.9 to 98.9] | 95.8 [93.2 to 97.6] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  H3N2: Day 1(N=606,705,306,358,NA,NA) | 77.6 [74.0 to 80.8] | 89.2 [86.7 to 91.4] | 80.4 [75.5 to 84.7] | 88.0 [84.2 to 91.2] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  H3N2: Day 22(N=606,705,306,358,NA,NA) | 98.7 [97.4 to 99.4] | 98.3 [97.0 to 99.1] | 99.0 [97.2 to 99.8] | 98.3 [96.4 to 99.4] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B1: Day 1(N=606,705,306,358,NA,NA) | 65.5 [61.6 to 69.3] | 70.9 [67.4 to 74.3] | 62.4 [56.7 to 67.9] | 67.9 [62.8 to 72.7] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B1: Day 22(N=606,705,306,358,NA,NA) | 96.4 [94.6 to 97.7] | 91.8 [89.5 to 93.7] | 96.4 [93.7 to 98.2] | 87.7 [83.9 to 90.9] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized
  B2: Day 1(N=606,705,NA,NA,297,361) | 73.8 [70.1 to 77.2] | 81.7 [78.6 to 84.5] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized | 72.7 [67.3 to 77.7] | 80.9 [76.4 to 84.8]
  B2: Day 22(N=606,705,NA,NA,297,361) | 99.3 [98.3 to 99.8] | 96.2 [94.5 to 97.5] | NA [NA to NA] — antigen not immunized | NA [NA to NA] — antigen not immunized | 99.0 [97.1 to 99.8] | 95.3 [92.6 to 97.2]

8. Secondary Outcome: 8.Geometric Mean Titres (GMT) in Subjects After Receiving One Dose of Either QIVc, TIV1c Against B2 Strain
Description: Immunogenicity of QIVc to TIV1c was assessed by GMT in subjects measured by HI assay, three weeks after vaccination with one dose of either QIVc or TIV1c.
  Superiority was established if the upper bound of the two-sided 95% CI for the ratio of GMTs (GMT TIV1c /GMT QIVc) for HI antibody does not exceed the superiority margin of 1.
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | QIVc (≥18 Years) | TIV1c (≥18 Years)
Number analyzed (Participants) | 1311 | 664
Titers
  Day 1(N=1311,664) | 45.9 [43.3 to 48.8] | 55.7 [51.6 to 60.2]
  Day 22(N=1311,664) | 135.4 [127.6 to 143.7] | 91.7 [85.7 to 98.2]
Statistical Analysis 1: Comparison: QIVc (≥18 Years) vs TIV1c (≥18 Years); Superiority of immune responses of QIVc to TIV1c in terms of ratios of GMT against influenza strain B2; Test type: Non-Inferiority or Equivalence — The upper bound of the 2-sided 95% CI for the ratio of GMTs (GMT TIV1c or TIV2c /GMT QIVc) for HI antibody should not exceed the superiority margin of 1; Ratios of GMT = 0.6, 95% CI 2-sided [0.6 to 0.7]

9. Secondary Outcome: 9.Percentages of Subjects Achieving Seroconversion After One Dose of Either QIVc, TIV1c Against B2 Strain
Description: Immunogenicity of QIVc to TIV1c was assessed in terms of percentages of subjects showing seroconversion or significant increase in HI antibody titers, against influenza strain B2, three weeks (day 22) after vaccination with QIVc or TIV1c Superiority was established if the upper bound of the two-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV1c - % seroconversion QIVc) for HI antibody in ≥ 18 years age group does not exceed the margin of 0 points
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥18 Years) | TIV1c (≥18 Years)
Number analyzed (Participants) | 1311 | 664
percentages of subjects | 36.6 [34.0 to 39.3] | 17.2 [14.4 to 20.3]
Statistical Analysis 1: Comparison: QIVc (≥18 Years) vs TIV1c (≥18 Years); Superiority of immune responses of QIVc to TIV1c in terms of seroconversion rates against influenza strain B2; Test type: Non-Inferiority or Equivalence — The upper bound of the 2-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV1c or TIV2c - % seroconversion QIVc) for HI antibody should not exceed the margin of 0 points; Difference between seroconversion rates = -19.4, 95% CI 2-sided [-23.2 to -15.5]

10. Secondary Outcome: 10.GMT in Subjects After Receiving One Dose of Either QIVc, TIV2c Against B1 Strain
Description: Immunogenicity of QIVc to TIV2c was assessed by GMT in subjects measured by HI assay, three weeks after vaccination with one dose of either QIVc or TIV2c.
  Superiority was established if the upper bound of the two-sided 95% CI for the ratio of GMTs (GMT TIV2c /GMT QIVc) for HI antibody does not exceed the superiority margin of 1
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | QIVc (≥18 Years) | TIV2c (≥18 Years)
Number analyzed (Participants) | 1311 | 658
Titers
  Day 1(N=1311,658) | 59.7 [56.4 to 63.0] | 43.8 [40.3 to 47.6]
  Day 22(N=1311,657) | 177.1 [167.8 to 187.1] | 76.3 [70.4 to 82.7]
Statistical Analysis 1: Comparison: QIVc (≥18 Years) vs TIV2c (≥18 Years); Superiority of immune responses of QIVc to TIV2c in terms of ratios of GMT against influenza strain B1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; Ratios of GMT = 0.5, 95% CI 2-sided [0.5 to 0.5]

11. Secondary Outcome: 11.Percentages of Subjects Achieving Seroconversion After One Dose of Either QIVc, TIV2c Against B1 Strain
Description: Immunogenicity of QIVc to TIV2c in terms of percentages of subjects showing seroconversion or significant increase in HI antibody titers, against influenza strain B1, three weeks (day 22) after vaccination with QIVc or TIV2c Superiority was established if the upper bound of the two-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV2c - % seroconversion QIVc) for HI antibody in ≥ 18 years age group does not exceed the margin of 0 points
Time Frame: Three weeks post vaccination (Day 22)
Population: Analysis was done on FAS population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥18 Years) | TIV2c (≥18 Years)
Number analyzed (Participants) | 1311 | 657
percentages of subjects | 39.7 [37.0 to 42.4] | 18.0 [15.1 to 21.1]
Statistical Analysis 1: Comparison: QIVc (≥18 Years) vs TIV2c (≥18 Years); Superiority of immune responses of QIVc to TIV2c in terms of seroconversion rates against influenza strain B1; Test type: Non-Inferiority or Equivalence — The upper bound of the 2-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV1c or TIV2c - %seroconversion QIVc) for HI antibody should not exceed the margin of 0 points; Difference between seroconversion rates = -21.7, 95% CI 2-sided [-25.5 to -17.7]

12. Secondary Outcome: 12.Number of Subjects Reporting Solicited Adverse Events (AEs) After One Dose of Either QIVc, TIV1c or TIV2c by Overall Age Group
Description: Safety was assessed in terms of number (%) of subjects reporting solicited local and systemic reactions, day 1 to 7 after vaccination with one dose of either four (4) strain inactivated quadrivalent cell based influenza vaccine (QIVc) or trivalent inactivated influenza vaccine (TIV1c or TIV2c)
Time Frame: Day 1 to 7 post vaccination
Population: Analysis was done on solicited safety data set i.e. all subjects in the exposed set with solicited adverse event data
Measure: Number; unit: Subjects
Arm/Group | QIVc (≥18 Years) | TIV1c (≥18 Years) | TIV2c (≥18 Years)
Number analyzed (Participants) | 1319 | 670 | 663
Subjects
  Any local | 551 | 240 | 242
  Injection site induration(hardness) | 134 | 55 | 60
  Injection site erythema (redness) | 167 | 80 | 68
  Injection site ecchymosis(bruising) | 56 | 26 | 35
  Injection site pain | 443 | 186 | 195
  Any systemic | 376 | 192 | 194
  Chills | 70 | 35 | 36
  Nausea | 89 | 38 | 43
  Myalgia | 156 | 80 | 77
  Arthralgia | 90 | 44 | 54
  Headache | 185 | 90 | 89
  Fatigue | 178 | 109 | 81
  Vomiting | 23 | 6 | 5
  Diarrhea | 77 | 42 | 42
  Loss of appetite | 81 | 45 | 39
  Any other | 66 | 20 | 30
  Use of analgesics / antipyretics for prophylasis | 6 | 2 | 1
  Use of analgesics / antipyretics for treatment | 8 | 2 | 3
  Body temperature | 7 | 5 | 3

13. Secondary Outcome: 13.Number of Subjects Reporting Unsolicited Adverse Events (AEs) After One Dose of Either QIVc, TIV1c or TIV2c by Overall Age Group
Description: Safety was assessed in terms of number (%) of subjects reporting unsolicited AEs (day 1 to 22 after vaccination), serious adverse events (SAEs), medically attended AEs, AEs leading to withdrawal from the study, new onset of chronic diseases (NOCDs), and concomitant medications (day 1 to day 181 post vaccination) after receiving one dose of either four (4) strain inactivated quadrivalent cell based influenza vaccine (QIVc) or trivalent inactivated influenza vaccine (TIV1c or TIV2c)
Time Frame: Day 1 to 181 post vaccination
Population: Analysis was done on unsolicited safety data set i.e. all subjects in the exposed set with unsolicited adverse event data
Measure: Number; unit: Subjects
Arm/Group | QIVc (≥18 Years) | TIV1c (≥18 Years) | TIV2c (≥18 Years)
Number analyzed (Participants) | 1324 | 673 | 665
Subjects
  Any AE | 213 | 99 | 110
  Any possibly related AE | 57 | 22 | 30
  SAE | 52 | 22 | 21
  Possibly/probably related SAE | 0 | 0 | 0
  AE leading to study withdrawal | 2 | 1 | 1
  Medically attended AE | 344 | 172 | 166
  NOCD | 62 | 25 | 29
  Death(N=1355,676,669) | 5 | 5 | 2

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from day 1to day 7 post vaccination, unsolicited AEs were collected from day 1 to day 22 post vaccination and SAEs were collected from day 1 to day 181
Description: All the unsolicited AEs were reported by non-systematic assessment and the solicited AEs were reported by systemic assessment.
  For SAEs- analysis was done on Unsolicited safety set. For Other Aes-analysis was done on overall safety set.
Groups:
- TIV1c (≥ 18 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV1c (H1N1, H3N2, B1) recommended for 2013-2014 season
- Total: Total Number of Subjects
Arm/Group | QIVc (≥18 Years) | TIV1c (≥ 18 Years) | TIV2c (≥18 Years) | Total
Serious Adverse Events (participants affected / at risk) | 52/1324 | 22/673 | 21/665 | 95/2662
Other Adverse Events (participants affected / at risk) | 681/1324 | 332/673 | 335/665 | 1348/2662
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QIVc (≥18 Years) (N=1324) | TIV1c (≥ 18 Years) (N=673) | TIV2c (≥18 Years) (N=665) | Total (N=2662)
HISTIOCYTOSIS HAEMATOPHAGIC (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0 | 1
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 | 1 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 1 | 1 | 5
CARDIAC ARREST (Cardiac disorders) | 0 | 2 | 1 | 3
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 5 | 0 | 2 | 7
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 | 2 | 1 | 5
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 | 0 | 1 | 5
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 1 | 0 | 2
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 2 | 2
CHEST DISCOMFORT (General disorders) | 0 | 0 | 1 | 1
CHEST PAIN (General disorders) | 1 | 0 | 0 | 1
CORONARY ARTERY RESTENOSIS (General disorders) | 0 | 0 | 1 | 1
DEATH (General disorders) | 0 | 1 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 1 | 0 | 2
STRANGULATED HERNIA (General disorders) | 1 | 0 | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 1 | 1
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 3 | 1 | 0 | 4
DIVERTICULITIS (Infections and infestations) | 2 | 0 | 0 | 2
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0 | 1
MENINGITIS VIRAL (Infections and infestations) | 1 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 0 | 3 | 5
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 | 0 | 1 | 1
PYELONEPHRITIS (Infections and infestations) | 2 | 0 | 0 | 2
SEPSIS (Infections and infestations) | 1 | 1 | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 1 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 1
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 | 1 | 1 | 2
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 1
ALCOHOLISM (Psychiatric disorders) | 0 | 1 | 0 | 1
BIPOLAR DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 2 | 0 | 0 | 2
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
IMPLANTABLE DEFIBRILLATOR INSERTION (Surgical and medical procedures) | 0 | 0 | 1 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 0 | 1 | 1
HYPERTENSION (Vascular disorders) | 2 | 0 | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QIVc (≥18 Years) (N=1324) | TIV1c (≥ 18 Years) (N=673) | TIV2c (≥18 Years) (N=665) | Total (N=2662)
DIARRHOEA (Gastrointestinal disorders) | 91 | 49 | 48 | 188
NAUSEA (Gastrointestinal disorders) | 96 | 39 | 46 | 181
CHILLS (General disorders) | 72 | 35 | 37 | 144
FATIGUE (General disorders) | 183 | 113 | 81 | 377
INJECTION SITE ERYTHEMA (General disorders) | 167 | 80 | 68 | 315
INJECTION SITE HAEMORRHAGE (General disorders) | 56 | 26 | 35 | 117
INJECTION SITE INDURATION (General disorders) | 134 | 55 | 60 | 249
INJECTION SITE PAIN (General disorders) | 444 | 187 | 195 | 826
DECREASED APPETITE (Metabolism and nutrition disorders) | 82 | 45 | 40 | 167
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 98 | 56 | 58 | 212
MYALGIA (Musculoskeletal and connective tissue disorders) | 160 | 83 | 79 | 322
HEADACHE (Nervous system disorders) | 191 | 93 | 93 | 377

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial